CLINICAL TRIAL: NCT07016230
Title: Phase 2, Multicenter, Open Label, Platform Study Investigating Tarlatamab (AMG 757) in Patients With Metastatic/Locally Advanced Small-Cell Lung Cancer (SCLC) and Other Poorly Differentiated Neuroendocrine Carcinomas (NECs), With Biomarker Analysis to Characterize Response/Resistance
Brief Title: Study Investigating Tarlatamab (AMG 757) in Patients With Metastatic/Locally Advanced Small-Cell Lung Cancer (SCLC) and Other Poorly Differentiated Neuroendocrine Carcinomas (NECs), With Biomarker Analysis to Characterize Response/Resistance (UNLOCK TARLATAMAB)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-515847-47-00; 2024/4014 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2025-05-16; First posted 2025-06-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Metastatic/Locally Advanced Small-Cell Lung Cancer; Metastatic/Locally Advanced Poorly Differentiated NEC; Metastatic/Locally Advanced High-grade MTC
Keywords: Metastatic/Locally Advanced Poorly Differentiated Neuroendocrine Carcinomas; Metastatic/Locally Advanced Small-Cell Lung Cancer (SCLC); TARLATAMAB; metastatic/locally advanced high-grade medullary thyroid carcinoma
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): patients with metastatic/locally advanced SCLC with any level of DLL3 expression
  Interventions: Drug: Tarlatamab
- Cohort 2 (Experimental): patients with metastatic/locally advanced other poorly differentiated NECs whatever the primary or high grade medullary thyroid carcinoma (MTC, capped at 4 patients) DLL3 positive by immunohistochemistry (IHC).
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — Patients enrolled in both cohorts will receive treatment with tarlatamab at the dose of 1 mg on D1, 10 mg on D8 and D15 and Q2W thereafter in a 28-day cycle. Tarlatamab will be administrated in intravenous route until disease progression, unacceptable toxicity, or consent withdrawal.

SUMMARY:
UNLOCK TARLATAMAB is an open-label, single arm, multicenter, phase 2 platform study that aims to evaluate the mechanisms of action and resistance to tarlatamab in metastatic/locally advanced Small-Cell Lung Cancer (SCLC) with any level of DLL3 expression and in other poorly differentiated Neuroendocrine Carcinomas (NECs) DLL3 positive. The two cohorts of patients are the following: i. cohort 1: patients with SCLC with any level of DLL3 expression. ii. cohort 2: patients with other poorly differentiated NECs whatever the primary or high grade medullary thyroid carcinoma (MTC, capped at 4 patients) DLL3 positive by immunohistochemistry (IHC). Patients enrolled in both cohorts will receive treatment with tarlatamab at the dose of 1 mg on D1, 10 mg on D8 and D15 and Q2W thereafter in a 28-day cycle. Tarlatamab will be administrated in intravenous route until disease progression, unacceptable toxicity, or consent withdrawal. Tumor and blood samples will be collected at baseline, on-treatment and at progression in order to identify biomarkers of drug response

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients with histologically confirmed diagnosis of metastatic/locally advanced SCLC with any level of DLL3 expression (Cohort 1) or other poorly differentiated NECs whatever the primary or high-grade MTC (Cohort 2) based on the most recent biopsy of a metastatic site. Tumors from Cohort 2 must be DLL3 positive defined as DLL3 ≥1% or H-score ≥1 by IHC
3. For patients with poorly differentiated NECs whatever the primary, the biopsy of the disease diagnosis should be reviewed by an expert pathologist. Large cell, small cell or not otherwise specified are eligible. In addition, the tumor must have a Ki67 >20% or mitotic rate >20 per 10 high-power fields. For prostate cancer, the diagnosis of NEPC must be based on phenotype analysis, which may include IHC markers such as neuron-specific enolase (NSE), Chromogranin A or CD56 in the majority of the tumor sample, or molecular alterations such as TP53, Rb1, and PTEN
4. High-grade MTC should be defined according to international medullary cancer grading system (IMCGS)
5. Patients with metastatic/locally advanced SCLC and other poorly differentiated NECs must have been treated with at least 1 line of prior therapy, including a platinum-based regimen (resistant or sensitive to platinum), have experienced progression on standard treatment, as determined by the investigator. Prior treatment with PD-(L) 1 inhibitors is allowed Specific cases: Patients with NEPC must have received at least 1 line of prior therapy, including a platinum containing regimen for de novo NEPC or an androgen signaling inhibitor (eg. abiraterone, enzalutamide, darolutamide and/or apalutamide) if treatment-emergent NEPC. Patients with high-grade MTC (capped at 4 patients) must have been treated with at least 1 prior therapy including a RET selective inhibitor if the presence of a RET mutation
6. Patients with NEPC and without a history of bilateral orchiectomy are required to remain on luteinizing hormone-releasing hormone (LHRH) analogue therapy during the course of protocol therapy
7. Patients must have an ECOG performance status ≤2 at the time of screening
8. Patients must have a minimum life expectancy of 3 months
9. Patients must have at least one radiologically measurable lesion according to response evaluation criteria in solid tumors (RECIST) v1.1 criteria
10. Patients must have a tumor site easily accessible to biopsy, avoiding bone biopsy when possible. Patient must have accepted to perform pre-treatment, on-treatment, and end-of-treatment tumor and blood biopsies
11. Patients must have adequate bone marrow reserve and organ function, based on local laboratory data within 21 days prior to cycle 1, day 1 defined as:

    * Platelet count ≥100 000/mm3 or ≥100 × 109/L (platelet transfusions are not allowed up to 14 days prior to cycle 1 Day 1 to meet eligibility)
    * Hemoglobin (Hgb) ≥9.0 g/dL (transfusion and/or growth factor support is allowed)
    * Absolute neutrophil count (ANC) ≥1500/mm3 or ≥1.5 × 109/L (use of growth factors is not allowed in the 14 days prior cycle 1)
    * Creatinine clearance (CrCl): Creatinine clearance (CrCl) ≥30 mL/min as calculated using the Cockcroft-Gault equation or measured CrCl; confirmation of CrCl is only required when SCr is >1.5 × ULN
    * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) and alkaline phosphatase (ALP) <3 x ULN (or <5 x ULN for patients with liver metastases)
    * Total bilirubin (TBL) <.5 x ULN (<3 x ULN in the presence of documented Gilbert's Syndrome [unconjugated hyperbilirubinemia]) or <2 X ULN for patients with liver metastases
    * Serum albumin ≥2.5 g/dL
    * Prothrombin time (PT) or Prothrombin time- international normalized ratio (PT-INR) and activated partial thromboplastin time (aPTT)/partial thromboplastin time (PTT)≤1.5 × (ULN), except for patients on coumarin-derivative anticoagulants or other similar anticoagulant therapy, who must have PT-INR within therapeutic range as deemed appropriate by the Investigator
12. Patients must have baseline oxygen saturation > 90% on room air
13. Females of reproductive/childbearing potential must have a negative serum pregnancy test at screening and must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and for at least 60 days for females after the last dose of study drug.

    Note : Methods considered as highly effective methods of contraception include:
    1. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

       * Oral
       * Intravaginal
       * Transdermal
    2. Progestogen-only hormonal contraception associated with inhibition of ovulation:

       * Oral
       * Injectable
       * Implantable
    3. Intrauterine device (IUD)
    4. Intrauterine hormone-releasing system (IUS)
    5. Bilateral tubal occlusion
    6. Vasectomized partner
    7. Complete sexual abstinence defined as refraining from heterosexual intercourse during and upon completion of the study and for at least 7 months for females after the last dose of study drug. Periodic abstinence (calendar, symptothermal, post-ovulation methods) is not an acceptable method of contraception
14. Female patients must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 60 days after the final study drug administration
15. Male patients must be surgically sterile or must withhold heterosexual intercourse or must be willing to use a highly effective birth control upon enrollment, during the treatment period, and for at least 60 days following the last dose of study drug
16. Male patients must not freeze or donate sperm starting at screening and throughout the study period, and at least 60 days after the final study drug administration
17. Patients must understand, sign and date the written informed consent from prior to any protocol-specific procedures performed. Patients should be able and willing to comply with study visits and procedures as per protocol
18. Patients must be affiliated to a Social Security System or beneficiary of the same

Exclusion Criteria:

1. Patients unwilling to participate to the biological investigations and to perform blood and tissue sample collection as required in the protocol
2. Patients with SCLC or other poorly differentiated NECs whatever the primary or high-grade MTC amenable for treatment with curative intent
3. Patients with well differentiated neuroendocrine tumors, whatever the grade, pheocromocytoma, paraganglyoma, or low grade MTC
4. Patients with evidence of interstitial lung disease (ILD) (including pulmonary fibrosis or radiation pneumonitis) or is suspected to have such disease by imaging during screening
5. Patients who experienced recurrent pneumonitis (grade 2 or higher) or severe, life-threatening immune-mediated AEs or infusion-related reactions including those that lead to permanent discontinuation while on treatment with immuno-oncology agents
6. Patients with a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients of tarlatamab
7. Inadequate washout period prior to cycle 1 day 1, defined as:

   1. Whole brain radiation therapy or stereotactic brain radiation therapy <14 days
   2. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation <28 days or palliative radiation therapy <7 days
   3. Any investigational agents or other anticancer drug(s) from a previous cancer treatment regimen or clinical study <30 days or < 5 half-lives, whichever is longer, prior to first dose of tarlatamab. Conventional chemotherapy eligible if at least 14 days or < 5 half-lives, whichever is longer, have elapsed and if all treatment-related toxicity has been resolved to grade ≤1
   4. Major surgery (excluding placement of vascular access) < 21 days
   5. Live virus and live-attenuated vaccination <28 days
   6. Systemic steroid therapy or other immunosuppressive therapy < 7 days
8. Prior treatment with tarlatamab or any selective inhibitor of the DLL3 pathway
9. Evidence of spinal cord compression or brain metastases, defined as being clinically active and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Patients with clinically inactive or treated brain metastases who are asymptomatic (ie, without neurologic signs or symptoms and do not require treatment with corticosteroids or anticonvulsants) may be included in the study. Patients must have a stable neurologic status for at least 2 weeks prior to cycle 1 day 1
10. Patients with evidence of any leptomeningeal disease
11. Patients with unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to grade 1 or baseline according to the NCI-CTCAE v5.0
12. Any evidence of primary malignancy other than metastatic/locally advanced SCLC, poorly differentiated NEC or high-grade MTC within 3 years prior to cycle 1 day 1, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated
13. Any evidence of severe or uncontrolled systemic diseases including active bleeding diatheses, active infection, psychiatric illness/social situations, geographical factors, substance abuse, or other factors which in the Investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardize compliance with the protocol. Screening for chronic conditions is not required
14. Patients with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of study treatment.
15. Patients with clinically significant pleural effusion will be excluded. Pleural effusion managed with indwelling pleural catheter (eg, PleurX) are allowed
16. Uncontrolled or significant cardiovascular disease prior to cycle 1 day 1, including:

    1. Corrected QT interval >470 ms for females and >450 ms for males according to Fridericia's formula (QTcF) and assessed based on triplicate ECGs, approximately 1 minute apart
    2. LVEF <50% by either echocardiogram (ECHO) or multigated acquisition (MUGA) scan
    3. Myocardial infarction within 6 months
    4. NYHA > class II within 6 months
    5. Clinically significant pericardial effusion as determined by an ECHO or MUGA scan
17. Patient with history of arterial thrombosis (eg, stroke or transient ischemic attack) within 12 months of first dose of tarlatamab
18. Active Hepatitis B and/or Hepatitis C infection, such as those with serologic evidence of viral infection within 28 days of cycle 1, day 1.

    Patients with past or resolved Hepatitis B virus (HBV) infection are eligible if:
    1. Hepatitis surface antigen (HBsAg) negative and hepatitis B core antibody (anti-HBc) positive; OR
    2. HBsAg positive and HBV deoxyribonucleic acid (DNA) viral load is documented to be ≤ 2000 IU/mL in the absence of anti-viral therapy and during the previous 12 weeks prior to the viral load evaluation with normal transaminases; OR
    3. HBsAg positive and HBV DNA viral load is documented to be ≤ 2000 IU/mL in the absence of anti-viral therapy and during the previous 12 weeks prior to the viral load evaluation with abnormal transaminases AST/ALT < 3 ULN.

    Patients with a history of Hepatitis C infection will be eligible for enrollment only if the viral load according to local standards of detection, is documented to be below the level of detection in the absence of anti-viral therapy during the previous 12 weeks (ie, sustained viral response according to the local product label but no less than 12 weeks, whichever is longer).
19. Patients with history or evidence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. Patient is eligible if no acute symptoms of coronavirus disease 2019 (COVID-19) within 14 days prior to first dose of tarlatamab (counted from day of positive test for asymptomatic subjects)
20. Patient with active or prior documented autoimmune or inflammatory disorders, including but not limited to inflammatory bowel disease [e.g. colitis or Crohn's disease], diverticulitis with the exception of diverticulosis, celiac disease or other serious gastrointestinal chronic conditions associated with diarrhea, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangitis), rheumatoid arthritis, hypophysitis, uveitis within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

    1. Patient with auto-immune alopecia
    2. Patient with Grave's disease, vitiligo or psoriasis not requiring systemic treatment within the last 2 years
    3. Patient with hypothyroidism (e.g. following Hashimoto syndrome) stable on thyroid hormone replacement
21. Patient with diagnosis of human immunodeficiency virus (HIV). Patients with HIV infection on antiviral therapy and undetectable viral load are allowed with a requirement for regular monitoring for reactivation for the duration of treatment on study per local or institutional guidelines
22. Female patients who are pregnant or breastfeeding or intend to become pregnant during the study
23. Patients with any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
24. Patients under guardianship or deprived of his/her liberty by a judicial or administrative decision or incapable of giving his/her consent
25. Prior history of severe or life-threatening events from any immune-mediated therapy
26. Participation in another clinical trial (<30 days or < 5 half-lives, whichever is longer) evaluating an experimental drug (except non-interventional research)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
To estimate the objective response rate (ORR) | Within the 4 months of treatment initiation

SECONDARY OUTCOMES:
Objective response rate at different timepoints (ORR) | up to 18 months
Duration of response (DOR) | From cycle 3 (Week 6; each cycle is 28 days) up to 2 years after the EoT, an average of 26 months
  defined as the time from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of progression (PD) or death due to any cause. Duration of response will be measured for responding patients (CR or PR) only
Clinical benefit rate (CBR) | During treatment period, a median of 4 months
  defined as the presence of at least a PR or CR, or a stable disease (SD) >6 months
Progression free survival (PFS) | From the time date of the first dose until progression or death from any cause, whichever occurs first, assessed up to 18 months
  defined as the time from date of first dose until the date of the first objective documentation of disease progression or death from any cause, whichever occurs first. For patients without documented radiological progression, follow-up will be censored at the date of last radiological assessment without progression, unless death occurs within 12 weeks following the date of last known progression-free, in which case the death will be counted as a PFS event
Frequency of all adverse events | From enrollment until 24 months of EoT
Severity of all adverse events | From enrollment until 24 months of EoT
  As defined by the NCI-CTCAE v5.0.
frequency of CRS and ICANS | From enrollment until 24 months of EoT
  graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria
severity of CRS and ICANS | From enrollment until 24 months of EoT
  graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria
Proportion of treatment discontinuation due to any AEs | Treatment Period, median of 4 months
Proportion of treatment interruptions due to any AEs. | Treatment Period, median of 4 months
Proportion of dose reductions due to any AEs | Treatment Period, median of 4 months
Severity of laboratory abnormalities | From enrollment until 24 months of EoT
  Defined by NCI-CTCAE v5.0
Frequency of laboratory abnormalities | From enrollment until 24 months of EoT

OTHER OUTCOMES:
mechanisms of action of tarlatamab | from enrollment unti EoT, with a median of 4 months
mechanisms of resistance of tarlatamab | from enrollment unti EoT, with a median of 4 months
Description of patient-reported outcomes (PROs) | Treatment Period, median of 4 months
  physical functioning sub-scale score of the EORTC QLQ-C30
Description of patient-reported outcomes (PROs) | Treatment Period, median of 4 months
  QoL scale score of the EORTC QLQ-LC13

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France